CLINICAL TRIAL: NCT05200637
Title: A Randomized, Parallel, Active Controlled Study to Evaluate the Vascular Response of Orsiro vs. Xience Drug Eluting Stent System in Subjects With Coronary Bifurcation Lesions
Brief Title: Vascular Response of Orsiro vs. Xience Drug-Eluting Stents for Treating Coronary Bifurcation Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ying-Chang Tung, Assistant Professor, Department of Cardiology, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202101599A3
Record Dates: First submitted 2022-01-04; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting stents; Coronary bifurcation lesions; Double-kissing crush technique; Optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients with true coronary bifurcation lesions will be randomized to undergo two-stent DK-crush technique with Orsiro or Xience. Another parallel prospective registry will enroll patients with bifurcation lesions treated with provisional one-stent strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Orsiro (Active Comparator): Two-stent DK-crush technique with Orsiro
  Interventions: Device: Orsiro stent
- Xience (Active Comparator): Two-stent DK-crush technique with Xience
  Interventions: Device: Xience stent
- Single stent (Other): Provisional one-stent strategy with any drug-eluting stent
  Interventions: Device: Any drug-eluting stent

INTERVENTIONS:
Device: Orsiro stent — Orsiro stent
  Arms: Orsiro
Device: Xience stent — Xience stent
  Arms: Xience
Device: Any drug-eluting stent — Any drug-eluting stent
  Arms: Single stent

SUMMARY:
This study aims to compare vessel response and clinical outcomes of a biodegradable-polymer, ultra-thin strut, drug-eluting stent (Orsiro, Biotronik) and a durable-polymer, thin-strut, drug-eluting stent (Xience, Abbott) for the treatment of coronary bifurcation lesions with two-stent double-kissing crush technique. How the differences in stent platforms affect vessel healing process will be examined by optical coherence tomography.

DETAILED DESCRIPTION:
Patients with true coronary bifurcation lesions (Medina [1, 1, 1] or [0, 1, 1]) will be enrolled and randomized to undergo two-stent double kissing crush technique with Orsiro or Xience. Pre-intervention and post-stenting optical coherence tomography will be performed during the index procedure. Another parallel prospective registry will enroll patients with bifurcation lesions treated with provisional one-stent strategy. All subjects will receive coronary angiography and optical coherence tomography follow-up at 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are at least 20 years old and present with acute or chronic coronary syndrome.
2. Patients who are suitable for PCI with DES implantation and provide written informed consent.
3. Patients with coronary bifurcation lesion amenable to be treated with 2-stent double-kissing (DK) crush technique.
4. Target vessels suitable for OCT examination.
5. Women of childbearing potential must have a negative pregnancy (serum and/or urine) test within 7 days prior to index procedure in accordance with the institutional standard of care. Female subjects who are surgically sterile or post-menopausal are exempt from having a pregnancy test.

Exclusion Criteria:

1. Patient who are not suitable candidates for use of dual antiplatelet therapy (DAPT)
2. Estimated glomerular filtration rate < 45 ml/min/1.73 m2
3. Liver cirrhosis
4. Life expectancy < 1 year
5. Planned surgery within 3 months
6. Pregnancy, breast-feeding, or plan to be pregnant in the coming 12 months
7. Target bifurcation lesion involved in chronic total occlusion or the culprit vessel of ST-elevation myocardial infarction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of stent strut coverage at bifurcation segments | 3 months post-procedure

SECONDARY OUTCOMES:
Neointimal thickness (μm) at bifurcation segments | 3 months post-procedure
Amount of in-stent intimal hyperplasia (mm3) at bifurcation segments | 3 months post-procedure
Amount of in-segment intimal hyperplasia (mm3) at bifurcation segments | 3 months post-procedure
Percentage of acquired malapposed struts at bifurcation segments | 3 months post-procedure
Percentage of stent strut coverage at bifurcation segments | 12 months post-procedure
Neointimal thickness (μm) at bifurcation segments | 12 months post-procedure
Amount of in-stent intimal hyperplasia (mm3) at bifurcation segments | 12 months post-procedure
Amount of in-segment intimal hyperplasia (mm3) at bifurcation segments | 12 months post-procedure
Percentage of acquired malapposed struts at bifurcation segments | 12 months post-procedure
In-stent late-lumen loss by quantitative coronary analysis | 3 months post-procedure
In-segment late lumen loss by quantitative coronary analysis | 3 months post-procedure
Target Lesion Revascularization (TLR) | 3 months post-procedure
Target Vessel Revascularization (TVR) | 3 months post-procedure
Target Lesion Failure (TLF) | 3 months post-procedure
  Cardiac death, target vessel related myocardial infarction (MI), and clinically indicated TLR
Major Cardiac Adverse Events (MACE) | 3 months post-procedure
  Cardiac death, myocardial infarction (Q wave and non-Q wave), emergent coronary artery bypass surgery, or target vessel revascularization (TVR)
Instent late-lumen loss by quantitative coronary analysis | 12 months post-procedure
In-segment late lumen loss by quantitative coronary analysis | 12 months post-procedure
Target Lesion Revascularization (TLR) | 12 months post-procedure
Target Vessel Revascularization (TVR) | 12 months post-procedure
Target Lesion Failure (TLF) | 12 months post-procedure
  Cardiac death, target vessel related myocardial infarction (MI), and clinically indicated TLR
Major Cardiac Adverse Events (MACE) | 12 months post-procedure
  Cardiac death, myocardial infarction (Q wave and non-Q wave), emergent coronary artery bypass surgery, or target vessel revascularization (TVR)
Stent thrombosis | 1 months post-procedure
  Stent thrombosis (all, definite, definite/probable, probable, possible) according to Academic Research Consortium (ARC) criteria for acute, subacute, late, very late and cumulative stent thrombosis
Stent thrombosis | 3 months post-procedure
  Stent thrombosis (all, definite, definite/probable, probable, possible) according to Academic Research Consortium (ARC) criteria for acute, subacute, late, very late and cumulative stent thrombosis
Stent thrombosis | 12 months post-procedure
  Stent thrombosis (all, definite, definite/probable, probable, possible) according to Academic Research Consortium (ARC) criteria for acute, subacute, late, very late and cumulative stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chang Tung, MD, Principal Investigator — Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan; Chi-Jen Chang, MD, Study Chair — Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan; Chia-Pin Lin, MD, Study Director — Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No